项目类别:

项目编号:

# 中山大学临床医学研究 5010 计划项目 任务书

项 目 名 称: 自体瘢痕真皮支架的组织工程皮肤移植修复增

生性瘢痕的多中心随机对照临床试验

承担单位: 中山大学附属第一医院

项目负责人: 吴军

联系电话: 02087755766-8235

手 机: 13983130289

电子邮箱: junwupro@126.com

起止时间: 2018年12月—— 2028年12月

# 填写说明

- 一、本任务书仅适用于我校满足相关条件的在编在岗教师填报项目 立项、实施及验收的基本依据。
- 二、填写任务书前,请先查阅《2. 中山大学高校基本科研业务费 专项资金实施试行办法》及《中山大学临床医学研究 5010 计划 纲要》。
- 三、本《任务书》各方可根据项目具体情况,就本《任务书》的未 尽事宜协商签订附加条款。附加条款与本《任务书》正文具有 同等法律效力。
- 四、《任务书》封面右上角请注明项目类别"常规"或"培育"。
- 五、本《任务书》中的表格如位置不够请自行加页。
- 六、《任务书》由申请人填写,经院系签署意见后,一式三份送科 学研究院。

一、项目基本信息

| I | 页目名称 | 自体癥 | 痕真皮 | | 工程皮肤移机对照临床 | 植修复增生性瘾<br>试验 | <b></b> 狼的多中心 |
|---|---|---|---|---|---|---|---|
| 项目 | 目承担单位 | 中山大学附属第一医院 | | | | | |
| 合作单 | 序号 | 单位名称 | | | | | |
| | 1 | | | 肇月 | 夫市第一人目 | 民医院 | |
| 位 | 2 | | | J- 3 | 东省工伤康复 | 省工伤康复医院 | |
| | 姓名 | | 吴军 | 2 | 性别 | 男 | |
| 项目 | 出生年月 | 1 | 962年 | 02 月 | 学历 | 博士研究生 | |
| 负 | 学位 | | 博士 | | 专业 | 创面修复,烧伤整形 | |
| 责人 | 职务 | | 学科带 | 头人 | 职称 | 教授 | |
| | 联系电话 | 13983130289 | | | E-mail | junwuproi | 0126.com |
| | 姓名 | 性别 | 年龄 | 职称 | 学历 | 单位 | 签名, つ |
| | 朱家源 | 男 | 56 岁 | 教授,主任<br>医师 | 博士研究生 | 中山大学附属第<br>一医院 | 2.2 |
| | 唐冰 | 男 | 47 岁 | 教授,主任<br>医师 | 博士研究生 | 中山大学附属第<br>一医院 | 1300 |
| | 胡志成 | 男 | 34 岁 | 副主任医师 | 博士研究生 | 中山大学附属第 一医院 | 胡玉净 |
| | 舒斌 | 男 | 43 岁 | 副主任医师 | 博士研究生 | 中山大学附属第 一医院 | Konsky |
| | 周强 | 男 | 48 岁 | 主任医师 | 博士研究生 | 肇庆市第一人民<br>医院 | 1274 |
| 主要 | 易先锋 | 男 | 56 岁 | 主任医师 | 博士研究生 | 广东省工伤康复 <sup>*</sup><br>医院 | 8233 |
| 参加人员 | 邹华春 | 男 | 38 岁 | 教授 | 博士研究生 | 中山大学公共卫<br>生学院(深圳) | 易好 |
| | 张利军 | 女 | 34 岁 | 博士后 | 博士研究生 | 中山大学附属第一医院 | 强利车 |
| | 刘旭盛 | 男 | 57 岁 | 教授,主任 医师 | 博士研究生 | 中山大学附属第一医院 | 2100 |
| | 谢举临 | 男 | 46 岁 | 教授,主任 医师 | 博士研究生 | 中山大学附属第一医院 | Sylm |
| | 徐盈斌 | 男 | 50 岁 | 主任医师 | 博士研究生 | 中山大学附属第一医院 | Hone |
| | 陈蕾 | 女 | 36 岁 | 副主任医师 | 博士研究生 | 中山大学附属第一医院 | 明温 |
| | 谢肖霞 | 女 | 43 岁 | 副主任护师 | 本科 | 中山大学附属第一医院 | 湖村村路 |
| | 梁月英 | 女 | 48 岁 | 副主任护师 | 本科 | 中山大学附属第一医院 | 2166 |

# 二、项目内容摘要及立项依据

#### 1、 项目内容摘要

增生性瘢痕是创伤修复的必然产物,其影响外观,部分瘢痕挛缩往往导致关节功能障碍。 患者生活质量低下,治疗周期长,社会负担重,医疗费用高。目前临床上植皮术是手术修复瘢痕的金标准。但是,往往存在皮源不足,易瘢痕复发,缺乏皮肤附属器官的问题。应用复合皮 移植方法,可减少瘢痕愈后复发的机率,缓解皮源不足。但是,其成活率不高,而且,脱细胞 异体真皮支架价格昂贵,医疗负担沉重。因此,如何有效修复手术切除瘢痕后的创面是亟需解 决的主要问题。

真皮缺失是瘢痕修复不满意和复发的主要原因。课题组前期的临床研究发现:应用术中实时快速获取的自体表皮基底细胞复合自体皮片移植治疗创面,能有效提高植皮成活率 (Brit J Surg, 2015)。进一步提出应用自体瘢痕真皮支架,可以实现取皮区损伤控制和自体瘢痕组织真皮支架的原位移植,有效降低了患者的经济负担。因此,我们猜想,如果用自体表皮基底细胞复合自体瘢痕真皮支架复合自体皮片,构建组织工程皮肤原位移植,修复瘢痕切除后创面,是否可以提高植皮成活率,减少瘢痕复发。为此,我们拟开展多中心、前瞻性随机对照临床试验,旨在对增生性瘢痕的修复提出更为有效的外科治疗指南,提高复合皮移植成活率,解决目前临床上增生性瘢痕修复的难题。

### 2、 立项依据(包括项目的意义和必要性、国内外现状和发展趋势)

### 课题研究的背景和必要性

增生性瘢痕是由于细胞异常增生以及细胞外基质沉积造成的皮肤纤维化异常,创伤修复的必然产物[1]。部位瘢痕突出皮面,形状不规则,高低不平,潮红充血,质地实韧。有灼痛和瘙痒感,于环境温度增高,情绪激动,或进食辛辣刺激性食物时症状加剧。增生往往延续几月或几年后才逐渐发生退行性变化,表现为突起高度减低,颜色转暗,充血消退,变软。有些最终可以平复,痛痒症状也大为减轻或消失。部分增生性瘢痕挛缩引往往导致关节功能障碍,影响外观和功能。大约 40%-70%的手术后以及 91%的烧伤后会形成增生性瘢痕[2]。据统计在美国每年至少 120 亿美元用于皮肤瘢痕的修复[3],给社会和经济带来巨大的负担。患者生活质量低下,治疗周期长,人力负担大,社会负担重,医疗费用高。

目前临床上植皮术是手术修复瘢痕的金标准。但是,往往存在皮源不足,易瘢痕复发,缺乏皮肤附属器官的问题。应用复合皮移植方法,可减少瘢痕愈后复发的机率,缓解皮源不足。但是,其成活率不高,而且,脱细胞异体真皮支架价格昂贵,医疗负担沉重。因此,如何有效修复手术切除瘢痕后的创面是亟需解决的主要问题。

真皮缺失是瘢痕修复不满意和复发的主要原因。课题组前期的临床研究发现:应用术中实时快速获取的自体表皮基底细胞复合皮片移植治疗创面,能有效改善植皮成活率(Brit J Surg, 2015)[4]。进一步应用自体瘢痕真皮支架,可以实现取皮区损伤控制和自体瘢痕组织真皮支架的原位移植,有效降低了患者的经济负担。因此,我们猜想,如果用自体表皮基底细胞复合自体瘢痕真皮支架复合自体皮片移植,修复瘢痕切除后创面,是否可以减少瘢痕复发,提高植皮成活率。为此,我们拟开展多中心、前瞻性随机对照临床试验,旨在对增生性瘢痕的修复提出更为有效的外科治疗指南,提高复合皮移植成活率,解决目前临床上增生性瘢痕修复的难题。

# 国内外的研究现状和发展趋势

组织工程学是 80 年代提出的一个崭新概念,融合了工程学和生命科学的基本原理、基本理论、基本技术和基本方法,在体外构建一个有生物活性的种植体,植入体内修复组织缺损,替代器官功能;或作为一种体外装置,暂时替代器官功能,达到提高生存质量,延长生命活动的目的。它的科学意义不仅在于为解除病人痛苦提供了一种新的治疗方法,更主要的是提出了复制"组织"、"器官"的新思想,它标志着"生物科技人体时代"的到来,是"再生医学的新时代",是"一场深远的医学革命"。组织工程的骨、神经、肌腱、软骨等都在进行着深入的研究,且取得了可喜的进展。与此同时,组织工程皮肤的研究也在不断的深入。

**组织工程皮肤**是指由细胞或细胞外基质或由两者共同结合组成的皮肤产品,是运用生命科学和工程学的原理与技术将种子细胞与适当的支架材料相结合构建出的用于修复、维护和改善损伤皮肤组织功能和形态的生物替代物。目前的组织工程皮肤包括组织工程表皮、组织工程真皮及组织工程复合皮3种。

组织工程表皮始于 1975 年 Rheinwald 和 Green[5]将表皮细胞在一层可供给营养物质的、经放射处理的 NIH/3T3 滋养层上进行培养,得到细胞的快速增殖,这一结果使体外大规模培养表皮细胞获得成功,从此以后,采用培养的表皮细胞膜片移植覆盖创面逐渐得到应用。美国Genzyme Tissue Repair 公司成功生产出自体表皮膜片(EpiceITM),主要用于治疗大面积烧烫伤病人。它是将病人自体的角质细胞在体外扩增培养后,移植到溃疡、大疙性表皮松懈症部位。培养自体表皮移植物的优点是提供了大量可供移植的表皮膜片或细胞,能迅速恢复皮肤的屏障作用,并获得良好的功能和美学效果。但是临床的实践发现,由于缺乏真皮结构的支持,表皮替代物在移植后存在疤痕增生严重,抗感染能力差,不耐磨,易破溃,弹性欠佳,柔软度差及移植后创面接受率低,易剥离脱落及形成水疱等缺点。

真皮替代物中代表性的有 Alloderm, Intega, oermagraft。Alloderm 是一种商品化的脱细胞 真皮基质,它保留了表皮层,基底膜可使角质形成细胞自由移动至支架材料,Kopp[6]经过对 67 例烧伤患者多中心对照实验证实, 该产品的应用效果相当于薄的自体刃厚移植物加上异体真 皮基质。Integra 是美国 Integra Life Sciences 公司生产的,用于早期创面的覆盖的异种来源的永 久性真皮替代物。它是戊二醛交联牛 [型胶原与 6-硫酸软骨素及氨基葡萄糖构成"真皮","表 皮"为硅橡胶薄膜,这种人工皮肤能诱发成纤维细胞长入及血管长入,且不易降解,在治疗大 面积烧伤创面有着明显的优势。由于 Integra 诱导再生的真皮组织具有典型的乳突状结构和网状 结构,而且愈合创面无瘢痕组织增生[7],所以在治疗瘢痕疙瘩和增生性瘢痕方面也具有显著的 效果。Dermagraft 是将新生儿包皮的成纤维细胞接种于可吸收聚乳酸纤维网上培养,成纤维细 胞在支架内增殖,分泌胶原、氨基多糖、生长因子等基质成分,成纤维细胞被埋在基质中,这 些细胞和胶原蛋白由内到外覆盖整个网架,构成人工真皮。Transcyte 以前称为 Dermagraft-TC, 是将新生儿的成纤维细胞接种于 Biobrane 上培养 4-6 周,形成与各含有高水平分泌的人基质蛋 白和大量生长因子的致密细胞组织。有研究表明它在异体移植中的粘附性与愈合度与自体移植 相当。修复裸鼠创面的实验结果证明,移植该组织工程化真皮 14 天后,裸鼠创面即已完全愈 合。但这种愈合仍然是靠创面四周的表皮增殖爬行至 Dermagraft 上面而实现的[8]。真皮替代物 虽然可以暂时覆盖创面但是由于缺少表皮,感染几率大大增加,且外观欠佳。理想的组织工程 化皮肤应该包括表皮层和真皮层。从而达到永久修复创面的目的。

Apligraf 是由 Bell 等人首先开发了的一种活性人皮肤替代物,即组织工程复合皮,类似

真正的皮肤,是将新生儿成纤维细胞溶于牛胶原中塑形,再在其表面接种新生儿表皮角质形成细胞。它在组织学上类似人的皮肤,可以分泌基质蛋白和生长因子,有较好的临床接受率。临床已应用于慢性静脉性溃疡[9]、糖尿病足溃疡[10]、烧伤[11-12]、外科急性创面[13-19]等多种皮肤缺损病例,并取得了良好效果。但是 Apligraf 用的细胞仍然是异体的,美国 FDA 批准该产品的适应症是慢性皮肤溃疡,也就是说靠 APligraf 内的成纤维细胞和表皮细胞分泌的生长因子和良好的覆盖促进创面愈合,仍然没有解决异体来源细胞抗原性的问题,不是一种永久性的皮肤替代物。而且,国外的这些组织组织工程皮肤替代物因为生产成本较高,价格昂贵,国内市场的推广和应用受到极大限制。

综上所述,尽管上述产品已在临床上应用,但是,仍存在较多的问题,与理想的组织工程 皮肤还有相当的差距。例如细胞培养周期长,有的覆盖物薄而易碎,有的创面愈合后瘢痕挛缩 明显,易破溃,抗感染能力差,组织工程构建的"皮肤"仍不具备完整的皮肤结构,缺乏毛囊、 汗腺等附属器结构等一系列的问题,使组织工程创面覆盖物还需进一步的改进和完善。

理想的组织工程皮肤替代物应当是具有正常皮肤的物征与功能,而目前最佳的替代物仍然是自体表皮替代物,因为其余的各种方法大多数仅显效于慢性溃疡和烧伤的患者,同时它们也都不同程度的存在切取困难、易于感染、免疫排斥和过敏等。培养表皮片由于缺乏真皮成分的支持,对机械损伤高度敏感,移植后易形成创面收缩和瘢痕增生,而且由于缺乏真皮,没有实现真正的皮肤重建。真皮替代物由于缺乏表皮,无活细胞,易感染,移植后易降解、收缩,在创面边缘易形成瘢痕。因此,理想的人工皮肤应包含表皮和真皮两层结构并且应当最大限度的满足下列优点:①两者之间连接紧密;②具有柔韧性和一定的机械强度,移植到创面后很快即与创面良好贴附;③安全、不携带病毒;④表皮与真皮成分能尽快完成自身增殖、分化和功能成熟,形成更接近于生理的永久性的皮肤替代物等;⑤与生物体能很好地相容;⑥便于消毒、贮存和运输。

我们在修复皮肤缺损时,应用异体脱细胞真皮与自体薄皮片的复合皮移植积累的丰富的经验,取得了较好的临床效果[20-22]。但同时也存在着成活率未能达到理想的要求、成活后皮片质地、色泽及皮肤功能与正常皮肤仍有差距的问题。异源性皮肤组织工程支架不仅花费较高且存在免疫原性、单纯的刃厚皮移植术后部位瘢痕增生程度明显等。近期,我们将一种快速获得皮肤基底细胞悬液的方法应用于临床,该细胞悬液在促进创面愈合、提高皮片成活率、改善愈后皮肤色泽质地等方面都有良好的效果(Brit J Surg, 2015)。并且,进一步应用自体瘢痕真皮支架,可以实现取皮区损伤控制和自体瘢痕组织真皮支架的原位移植,有效降低了患者的经济负担,有效解决市场上脱细胞异体真皮支架价格昂贵等问题。因此,构成组织工程皮肤的两大要素已经齐备,我们拟将这两种技术结合在一起应用,得到一种快捷、有效的构建出有完整功能皮肤的方法,改善目前增生性瘢痕治疗的难题是本临床试验的目的。

#### 研究的目的和意义

综上所述,综合近年来的国内外研究进展,以及我们前期开展的临床研究结果,我们拟开展多中心,前瞻性、随机对照临床研究,将自体表皮基底细胞复合自体瘢痕真皮支架,结合自体皮片移植应用于增生性瘢痕的修复上,探索该方法的有效性和安全性。旨在为增生性瘢痕的治疗提出一个更为有效的外科治疗指南,提高植皮成活率,解决目前临床上的难题。从而提高患者生活质量,另外在缩短住院时间,减少患者治疗费用的同时,有效节约了医疗资源,具有极其重要的意义。

#### 参考文献:

- [1] Campaner AB, Ferreira LM, Gragnani A, et al. Upregulation of TGF- β1 expression may be necessary but is not sufficient for excessive scarring. J Invest Dermatol 2006; 126: 1168-1176.
- [2] Shi J, Shi S, Wu B,Zhang J,Li Y,Wu X,Zhang J,Wang K,Zhao B,Cai W,Bai X,Hu D,Guan H. Autophagy protein LC3 regulates the fibrosis of hypertrophic scar by controlling Bcl-xL in dermal fibroblasts. Oncotarget 2017;8(55):93757-70.
- [3] Finnerty CC, Jeschke MG, Branski LK, Barret JP, Dziewulski P, Herndon DN. Hypertrophic scarring: the greatest unmet challenge after burn injury. The Lancet 2016;388(10052):1427-36.
- [4] Hu ZC, Chen D, Guo D, Liang YY, Zhang J, Zhu JY, Tang B. Randomized clinical trial of autologous skin cell suspension combined with skin grafting for chronic wounds. Brit J Surg, 2015 Jan;102(2):e117-23.
- [5] Rheinwald JG, Green H. Serial cultivation of human epidermal keratinocytes: the formation of keratinizing colonies from single cells. Cell. 1975, 6(3):331-343.
- [6] Kopp J, Jeschke MG, Bach AD, et al. Applied tissue engineering in the closure of severe burns and chronic wounds using cultured human autologous keratinocytes in a natural fibrin matrix. Cell Tissue Bank. 2004;5(2):89-96.
- [7] Yannas IV. Studies on the biological activity of the dermal regeneration template. Wound Repair Regen. 1998, 6(6):518-523.
- [8] Hansbrough JF, Dore C, Hangsbrough WB. Clinical trial of a living dermal tissue replacement placed beneath meshed, split-thickness skin grafts on excised burn Wound. J Burn Care Rehabil 1992, 13(5):519-529.
- [9] Falanga V, Sabolinski M. A bilayered living skin construct (APLIGRAF) accelerates complete closure of hard to heal venous ulcers. Wound Repair Regen. 1999, (4):201-207.
- [10] Veves A, Falanga V, Armstrong DG, et al. Apligraf Diabetic Foot Ulcer Study Graftskin, a human skin equivalent, is effective in the management of noninfected neuropathic diabetic foot uleers: a Prospective randomized multicenter clinical trial. Diabetes Care, 2001, 24(2):290-295.
- [11] Waymack P, Duff RG, Sabolinski M. The effect of a tissue engineered bilayered living skir analog, over meshed split-thickness autografts on the healing of exeised burn Wounds- The Apligaf Burn Study Group. Burns, 2000, 26(7):609-619.
- [12] Hayes DW, Jr Webb GE, et al. Full-thickness burn of the foot: successful treatment with Apligraf A case report. Clin. Podiatr. Med. Surg. 2001,18(1):179-188.
- [13] Eaglstein WH, Alvarez OM, Auletta M, et al. Acute excisional wounds treated with a tissue engineered skin (Apligaf). Dermatol. Surg. 1999, 25(3):195-201.
- [14] Muhart M, MeFalls S, Kirsner R, et al. Bioengineered skin. Lancet, 1997, 350(9085):1142.
- [15] Muhart M, MeFalls S, Kirsner RS et al. Behavior of tissue-engineered skin: a comparison of a living skin equivalent, autograft, and occlusive dressing in human donor sites. Arch. Dermatol 1999, 135(8):913-918.
- [16] Eaglstein WH, Iriondo M, Laszlo K. A composite skin substitute (Graftskin) for surgical wounds. Dermatol. Surg. 1995, 21(10): 839-843.

- [17] Gohari S, Gambla C, Healey M, et al. Evaluation of tissue-engineered skin (human skir substitute) and secondary intention healing in the treatment of full thickness wounds after Mohs micrographic or excisional surgery. Dermatol Surg, 2002, 28(12): 1107-14, discussion 1114.
- [18] Tarlow MM, Nossa R, Speneer JM. Effective management of difficult surgical defects using tissue engineered skin. Dermatol. Surg.2001, 27(1):71-74.
- [19] Lee DK, and Serkin AL. Carbon dioxide laser and Apligraf for a painful plantar hypertrophic scar. J Am Podiatr Med Assoe.2004, 94(1):61-64.
- [20] Tang B, Zhu B, Zhu JY, et al. Early eschorectomy and concurrent composite skin grafting ovre human acellular dermal matrix scaffold for covering deep facial burns. Plast Reconstr Surg.2011. 127(4):1533-8.
- [21] 唐冰,朱家源,朱斌,等,复合皮混合移植治疗深 II 度烧伤创面的远期疗效观察.中山大学学报(医学科学版),2006(S2),27,192-194.
- [22] 朱家源,朱斌,李新强,等. 复合皮混合移植治疗深 II 度烧伤患者创面疗效观察. 中华烧伤杂志, 2005, 21(1): 21-23.

# 三、项目研究内容及预期目标

3、 研究目标(目标明确,请提出需要解决的具体临床问题)

通过采用多中心、前瞻性、随机对照临床研究,观察自体瘢痕真皮支架的组织工程皮肤移植修复增生性瘢痕(即以自体瘢痕作为真皮支架,同时结合术中实时快速获取的基底层细胞悬液作为种子细胞和自体皮片移植)有效性和安全性,恢复皮肤功能和改善质量,同时降低医疗费用。

#### 4、 研究内容

(1)有效性:通过多中心前瞻性随机对照临床试验,评价自体表皮基底细胞结合自体瘢痕真皮支架,复合自体皮片移植修复增生性瘢痕可以提高植皮成活率,其植皮成活率优于常规对照组。同时,评价植皮愈后效果(如术后瘢痕增生评分,色泽评分等),创面复发率。

(2)安全性:评价自体表皮基底细胞结合自体瘢痕真皮支架,复合自体皮片移植修复增生性瘢痕术后的并发症发生率,以及患者生活质量的差别。

- (3)评价医疗费用
- (4)评价随访期疗效
- 5、 研究方案及技术路线(包括研究的样本量、入选、排除、退出标准,研究结果的评价、知情同意、伦理学、质量控制等内容)

#### 1. 研究中心:

本研究为多中心、前瞻性、随机对照临床试验,研究单位有3个,中山大学附属第一医院烧伤科为牵头单位,肇庆市第一人民医院,广东省工伤康复医院为参与单位。

#### 2. 研究的持续时间和例数

本项临床试验计划拟于 2018 年 6 月开始,至 2027 年 12 月结束,整个研究过程为 10 年。本研究为多中心、前瞻性、随机对照临床试验。目标病例数为 226 例(具体样本量估算见后文)符合入选/排除标准的增生性瘢痕患者,每组 113 例。

### 3. 受试者的选择:

#### 3.1 入选标准

(1)受试者签署知情同意书当天的年龄为 0 天至 80 岁 364 天(如患者为未成年人,应由法定 监护人签署);

(2)诊断为增生性瘢痕,需行手术修复者;

- (3)瘢痕大小 10cm2-200cm2, 部位不限;
- (4)生命体征稳定,经常规检查表明可耐受手术者;(5)患者精神状态良好、能遵循医嘱,定期复诊者;
  - (6)研究人员认为不宜纳入者;
  - (7)患者在过去任何时间参加这项研究。

#### 3.3 剔除标准

对已被选入本临床研究,属于以下情况之一者,统计时作为剔除病例:

- (1)入选受试者后发现有不符合病例入选标准情况者;
- (2)入选后随访时间小于2次,而无法评价客观疗效者(但可评价不良反应);
- (3)违反试验方案要求的受试者。

#### 3.4 退出标准

受试者可以在任何时候、以任何理由退出临床试验。研究者认为不适宜继续治疗时从受试 者利益出发,也可要求受试者退出。

如果试验过程中受试者发生以下情况之一,研究者应当安排其中断治疗并退出试验:

- (1)受试者依从性差,不能遵循医嘱者;出现不良反应,研究者判断不宜继续进行本临床研究;受试者不愿意继续进行本临床研究自行退出。
- (2)退出试验前,必须完成最近一次随访及各项有关疗效和不良反应指标的评估,详细记录 退出病人的退出理由与日期。

#### 4. 研究过程

受试者入选后,按照随机分组的方法将受试者分配到试验组或对照组,在对临床试验进行 监查时须对受试者的入选、分组情况进行复核。

治疗方案:

#### 4.1 患者筛选期 (第-10 天至第 0 天内; 访视 1):

每位受试病人在进入试验之前必须完成下列项目,筛查结果在入组手术前10天内有效:

- ①签署知情同意书
- ②病史回顾
- ③个人基本资料
- ④常规体查,包括身高、体重和生命体征
- ⑤体格检查, 创面等专科检查
- ⑥血清/尿妊娠试验

#### 4.2 患者入组 (第1天; 访视2)

4.2.1 继续审查有否不良事件发生,如有需记录在病例记录表中。

#### 4.2.2 随机分组:

随机分配到试验组或对照组,按照瘢痕大小 10-50cm2, 50-200cm2 进行分层。由统计学专家应用 SAS 统计软件包随机分组,产生的随机分配序列,实时短信联系获取受试者随机入组类别。同时,随机分组信息由统计学专家备份保存。

受试者按照随机划分的组别,分别接受传统自体皮片移植手术(对照组)治疗和自体表皮基底细胞结合自体瘢痕真皮支架复合自体皮片移植手术(试验组)治疗(具体手术操作见下文4.2.1 手术实施方案)。

#### 4.2.1 手术实施方案:

- (1) 试验组手术方案:
- ① 瘢痕切除/削除,瘢痕中间真皮层予辊轴刀削除厚约 0.01-0.02mm 瘢痕组织,清洗干净后,予轧皮机轧制打孔拉网备用;
- ② 电动取皮刀取患者自体皮片,其中剪出一小块皮片(按取皮皮片与植皮创面大小比例为 1:80决定),按自体表皮基底细胞提取盒说明,配制成自体表皮基底细胞悬液备用;余下所取 皮片大小应为创面大小相当,生理盐水冲洗后,湿纱包裹备用。
- ③ 瘢痕切除创面将制备好的自体瘢痕真皮支架拉网移植于创面上,在网孔间及真皮支架上 喷洒或涂沫制备好的自体表皮基底细胞,自体皮片移植创面上,加压包扎固定:
  - ④ 术后按常规治疗定期更换外层敷料,按实验方案观察记录创面情况。
  - (2) 对照组手术方案:
  - ① 瘢痕切除/削除:
  - ② 自体皮片移植于创面上,加压包扎固定:
  - ③ 术后按常规治疗定期更换外层敷料,按实验方案观察记录创面情况。

#### 4.2.2 完成 CRF 表中手术记录。

#### 4.3 访视 3 (术后第 7±1 天)

- (1) 进行体格检查和记录生命体征,并记录在病例报告表上;
- (2) 审查和收集/记录受试者入组以来接受的所有联合用药。所有联合用药必须记录在适当的病例报告表上:
  - (3) 监测不良事件: 自手术后以来任何不良事件必须记录在适当的病例报告表上;
  - (4) 监测植皮区情况:关于植皮区访视情况的结果按要求记录在病例报告表上。

#### 4.4 访视 4 (术后第 14±2 天)

- (1) 进行创面检查和记录生命体征,并记录在病例报告表上;
- (2) 监测不良事件: 自手术后以来任何不良事件必须记录在适当的病例报告表上;
- (3) 监测植皮区情况: 收集植皮后创面信息,所有关于植皮区情况的结果必须记录在病例报告表上;

#### 4.5 访视 5 (术后第1月±5天)

- (1) 进行创面检查和记录生命体征,并记录在病例报告表上;
- (2) 监测不良事件: 自手术后以来任何不良事件必须记录在适当的病例报告表上;
- (3) 监测植皮区情况: 收集植皮后创面信息, 所有关于植皮区情况的结果必须记录在病例报告表上;

#### 4.6 访视 6 (术后第 3 月±7 天)

- (1) 进行创面检查和记录生命体征,并记录在病例报告表上;
- (2) 监测不良事件: 自手术后以来任何不良事件必须记录在适当的病例报告表上;
- (3) 监测植皮区情况: 收集植皮后创面信息, 所有关于植皮区情况的结果必须记录在病例报告表上;

#### 4.7 访视 7 (术后第 6 月 ± 7 天)

- (1) 进行创面检查和记录生命体征,并记录在病例报告表上;
- (2) 监测不良事件: 自手术后以来任何不良事件必须记录在适当的病例报告表上:
- (3) 监测植皮区情况: 收集植皮后创面信息, 所有关于植皮区情况的结果必须记录在病例报告表上;

#### 5. 疗效评价

#### 5.1 疗效评价标准

按植皮成活率(等同于创面愈合率)、国际通用的疼痛(VAS)评分、患者与温哥华瘢痕量表(VSS)等的疗效评价标准对植皮区进行评价。

#### 5.2 疗效评价指标

①瘢痕评分: 在术后 6 月时进行瘢痕评分,评价效果

- ②植皮成活率(创面愈合率): 在术后各个访视时间点对术区进行评估, 创面有否完全愈合;
- ③瘢痕复发率: 在术后 6 月时评价瘢痕复发率;
- ④VAS 疼痛评分: 在术后访视 3、4 时对术区进行评估疼痛(具体评分详见本章 14. 附件 1);
- ⑤温哥华瘢痕量表: 在术后各个访视时间点的术区进行评估瘢痕(具体评分详见本章 14. 附件 2)
  - ⑥发汗实验: 在术后 6 月时评价是否有发汗功能的恢复
  - ⑦毛发生长率: 在术后 6 月时评价毛发生长率

#### 5.3 疗效评价的时间

在本研究手术治疗后及后续随访中进行疗效评价,所有病人在完成或退出时均需进行疗效评估,之后进入随访期术后1周、2周、1个月、3个月、6个月、12个月各随访一次,并每次随访进行创面植皮术后评价。

#### 5.4 疗效评价的手段

为确保评价可靠,体表外观及功能要求两位医师(不知道受试者入选组别)体检进行评价 并如实记录于原始病历中作为客观证据。

#### 6. 安全性评价

所有在试验阶段发生的不良事件都应当记录,并由研究者判断和试验药物之间的因果关系。 任何在试验中出现且在试验结束时仍然异常的实验室检查结果,研究者应当追踪到这些指标恢 复正常或临床表现稳定为止。

#### 6.1 安全性指标

#### 6.1.1 生命体征和体格检查

在研究开始之前和受试者的每次访视时,必须记录下述的生命体征和体格检查结果。以下 是病人每次随访时必须检查的项目:

创面检查、心率、血压、体温、呼吸频率

#### 6.1.2 实验室检查指标

在开始研究之前,相应的临床监查员将记录参与实验室的正常值范围。在研究期间(访视1) 需要进行以下的实验室项目检查:

① 血清/尿妊娠试验(生育年龄女性需在访视1检查)

#### 6.1.2 安全性评价指标

不良反应, 如感染率、皮片坏死率、皮片坏死组织时, 皮片血管再生。

#### 6.2 不良事件评价

按不良事件评价表进行对照记录。

#### 7. 不良事件记录与报告

#### 7.1 定义

临床试验中的受试者在术后出现的任何非期望的和治疗有关或无关的医学事件都是不良事件。它可以是任何不利的和非期望的体征、症状、实验室检查等异常结果,而无论其是否和手术有关。所有的不良事件均应记录在 CRF 表中。

临床监查员在拜访研究中心时,必须在检查受试者的临床病历资料(原始数据核对)时系统性收集和核实关于不良事件的信息资料。需要继续随访在评估时还未解决的不良事件直至其解决。对于在临床可能的观察期间不能解决的不良事件(如截肢等),研究者将定级为永久性不能解决的事件,CRF 表中该事件解决的时间留空不填。

#### 7.2 不良事件相关性

研究者应对不良事件和手术以及合并用药之间可能存在的关联做出评估,参照以下 5 级分 类标准评定:

- (1) 肯定有关:反应出现符合手术后合理的时间顺序,反应符合所疑植皮手术已知的不良 反应类型。
- (2) 可能有关:反应出现符合手术后合理的时间顺序,反应符合所疑植皮手术已知的不良 反应类型;病人的临床状态或其他治疗方式也有可能产生该反应。
- (3) 可能无关:反应出现不太符合手术后合理的时间顺序,反应不太符合所疑植皮手术已知的不良反应类型;病人的临床状态或其他的治疗方式有可能产生该反应。
- (4) 无关:反应出现不符合手术后合理的时间顺序,反应有符合合并用药已知的反应类型,病人的临床状态或其他的治疗方式可能产生该反应,疾病状态改善或停止其他治疗方式反应消除,重复使用其它治疗方法反应出现。
- (5) 无法评定:反应出现与手术后的时间顺序无明确关系,与该植皮手术已知的不良反应 类型相似,同时使用的其他药物也可能引起相同的反应。

以上(1)、(2)、(5)项目记为本研究的不良反应。

不良反应发生率=不良反应例数/总例数×100%。

#### 7.3 不良事件分级标准

作为执业医师, 研究者将对所有不良事件进行如下评估:

(1) 轻度——意识到体征或症状,但容易耐受(对于儿科临床研究,定义为意识到症状,但容易耐受)

- (2) 中度——不适足以影响日常活动(对于儿科临床研究,定义为患儿的动作肯定有问题)
- (3) 重度——残疾,无法工作或进行日常活动(对于儿科临床研究,定义为极度痛苦或不能进行日常活动)

#### 7.4 严重不良事件

严重不良事件的定义为在手术后发生的非期望的不良事件,并符合以下标准中的任意一项: 1)导致死亡;2)由手术所致的危及生命;3)导致住院或延长住院时间;4)永久或显著丧失功能/残疾;5)致畸或致癌。

有些需要住院或延长住院时间的事件可不作为严重不良事件报告,包括:1)因社会原因而非不良事件住院;2)在进入研究前已经预约的择期手术,检查或其它治疗而住院。3)因已存在的并且没有在研究期间加重的疾病而住院。

#### 7.5 报告过程

#### 7.5.1 报告表

严重不良事件的报告需要使用 SAE 报告表。

#### 7.5.2 报告程序

严重不良事件的报告需要使用 SAE 报告表。出现严重不良事件时(与植皮手术相关或不相关),研究者应在 24 小时内将填写最初报告发送到中山大学附属第一医院伦理委员会(电话: 020-87755766-8185),并尽快将最终报告(包括严重不良事件转归等,如严重不良事件为死亡,则不必再追发最终报告)完成后再次报告上述部门。

#### 8. 退出和停止研究规则

#### 8.1 受试者退出

受试者可以在任何时候、以任何原因退出临床试验,而且不会影响研究者对其疾病治疗的权利。研究者从受试者的利益角度考虑,有权以任何理由包括伴发疾病、不良事件或治疗失败要求受试对象退出。临床研究核心小组保留由于方案违反、管理原因,或其它有效的和伦理性原因而要求受试对象退出的权利。

虽然应该尽可能的避免受试对象的退出,但是需要知道在临床研究中是会出现受试对象 退出的情况。不论受试对象在何时、以任何原因退出研究,必须完成该受试对象最后研究评估,并注明退出原因。有关该受试对象的所有文件资料都必须尽可能的完整。只要受试者没有撤回他的同意书,就要对这些退出受试者进行随访并且记录疾病情况,犹如他们没有退出一样。

研究者必须对由于依从性差而退出者进行跟踪随访以获得未参加随诊的原因。当病人退出,研究将应尽其所能尽可能全面地来完成和汇报观察到的资料。只要受试者没有撤回他的同意书,如果可能,将继续随访这些受试者并且记录疾病情况,犹如他们没有退出一样。

由于伴发疾病或不良事件而退出者,必须在观察表中详细记录,并附上所有其它适当的和 有价值的资料。

### 8.2 研究提前终止

提前终止的原因可包括外部事件、严重不良事件的重复发生、治疗相关的死亡率升高或临床试验的入组病例数不足。当提前终止临床研究时,所有研究者都将收到书面的通知。任何研究者如果想停止参与本项临床研究都必须将他/她的决定立即告知主要研究者。

### 8.3 研究的随访

8.3.1 随访时间

受试者在术后1周、2周、1月、3月、6月和12月各随访一次。

8.3.2 随访内容

受试者随访内容包括收集受试者一般生命征情况和创面检查,植皮区评价。将上述随访内容记录于原始病历中。评价内容需填写于 CRF 表中。

### 9. 统计学方法

### 9.1 样本量计算

本研究的初始评价指标为实验组的术后瘢痕评分优于对照组。

因此,研究假设1:

HO: 两组术后瘢痕评分相同

H1: 两组术后瘢痕评分不同

a = 0.05 (two sided)

$$n_1 = n_2 = 2 \left[ \frac{(z_{\alpha/2} + z_{\beta})\sigma}{\delta} \right]^2$$

我们取用优效性检验,假设对照组术后瘢痕评分为 12 分,实验组可提高 3 分,病人最长随访时间为 12 月,将采用双侧 0.05 显著性检验,20%的检验效能,从公式得出每组约需 96 例病人,考虑到受试者在 12 个月随访期内可能出现约 15%的脱失率,则每组约需 113 例病人,共需 226 例病人。考虑分层因素影响,该样本量也足够函括。

#### 9.2 主要终点指标

本研究的主要终点指标是术后6月瘢痕评分。

#### 9.3 次要终点指标

本研究的次要终点指标是术后 2 周植皮成活率(创面愈合率), VAS 疼痛得分, 植皮区色泽情况, 发汗功能, 毛发生长率, 不良反应率(如感染、皮片坏死等)。

#### 9.4 疗效

瘢痕评分:分析集受试者手术后术区(植皮区和供皮区)的瘢痕评分;

创面愈合率:分析集受试者手术后各随访点创面完全上皮化的病例数;

瘢痕复发率:分析集受试者手术后术区瘢痕复发情况;

温哥华量表得分:分析集受试者术区出现瘢痕增生的评分;

VAS 评分得分:分析集受试者术区感觉 VAS 评分得分;

发汗实验:分析集受试者术区发汗功能情况;

毛发生长率:分析集受试者术区毛发生长情况。

#### 9.5 安全性

在治疗过程中记录的实验室参数指标、症状和生命征指标。不良反应(包括植皮术区周围组织反应,有无充血、水肿、溃烂渗液等局部炎症反应或发热等全身反应征象,皮疹、搔痒及其它过敏现象,感染情况等),不良事件定义详见前述。

#### 9.6 分析

基线资料的均衡性分析通过频率列表进行描述性分析,采用卡方检验对两组基线资料进行比较。通过表格对两组之间每个相关特征的相似性进行分析。不对这些特征进行统计学假设检验。需要显示接受筛选、随机分组的受试者人数和百分比、筛选失败的主要原因以及停止治疗的主要原因。根据描述性统计值或分类表格按不同治疗组总结人口统计学变量(例如年龄、性别、人种)、主要和次要诊断、既往治疗和联合治疗。

#### 9.6.1 疗效

各疗效指标将以 95%可信区间来表示,将采用卡方检验、Fisher's 精确概率检验或 CMH 方法进行两组比较。使用 Miettinen 和 Nurminen 提议的方法,计算 95%置信区间。

## 9.6.2 有效性

分类数据如不良事件和严重不良事件将通过频率列表和总结图表来表现,将采用卡方检验、Fisher's 精确概率检验或 CMH 方法进行两组比较。

定量数据(如实验室检查)将应用算术平均数或中位数来描述其居中趋势,以及通过标准差或四分位间距来描述其分布范围,将采用 t 检验或非参数检验方法进行两组比较。

### 11.2 知情同意

受试者在入选试验前,研究者必须向他们解释试验目的,方法,可能的受益,潜在的风险和可能出现的不适。告知受试者参与试验是自愿的,可以在任何时候退出,是否参与试验对其疾病的治疗没有任何影响。受试者的隐私权将受到保护。

受试者或监护人员应有足够时间来阅读知情同意书和提出疑问。在入选前,受试者或其监护人必须签署知情同意书,受试者保留知情同意书的复印件。

# 11.3 临床研究管理规范 (GCP)

本临床研究将按照《赫尔辛基宣言》和中国临床研究管理规范(GCP)进行。本研究方案 必须经临床研究负责单位伦理委员会通过后方可实施。研究者将保证本临床研究遵守中华人 民共和国有关医学研究的法律、法规、科学和伦理标准来进行。若本研究方案在研究过程中 发现需要进行修订,修订的研究方案须再次报请负责单位伦理委员会备案/通过后方可实施。 如发现涉及研究药品的重要新资料,须将知情同意书作书面修改送负责单位伦理委员会通过, 并须再次取得受试者同意。

# 11.4 受试者个人资料的保密

本次试验中只收集局限于对植皮手术治疗的有效性、安全性等研究所需要的信息。收集和使用这些数据时将遵守相关的保护隐私权的法律和规定。

# 12. 管理要求和质量控制

## 12.1 方案的修改

研究者不能随意修改试验方案。如由于在试验过程中需要修改,所有的方案修改都将由 研究者向中山大学提出,经讨论同意后发布修改方案。

# 12.2 病例报告表的完成:

研究者首先按照"筛选表"的内容,确定受试者入组,入组后按方案要求进行检查及治疗,将有关内容记录于原始病历中,严格将原始病历及检查结果填写于 CRF 的"观察表"中,每一试验周期结束后填写"合并用药表"。研究结束后,填表医生/护士与上级医生一起认真复核 CRF 是否与原始记录一致。对显著偏离或在临床可接受的范围以外的数据必须加以核实,并由填表医生/护士和上级医生作必要说明。

# 12.3 数据质量保证

为了保证数据的完整性、准确性和可靠性,本次研究中采取了以下措施(另有 SOP 进一步详细规范本临床试验):

近期随访数据采用 Logistic 回归模型对相关预后因素进行分析,远期随访数据采用多因 素 Cox 回归模型对相关预后因素进行分析。

另外,缺失数据将采用末次观察结转法。

# 9.7 分析集的定义

分析集: ITT (intention to treat) 分析, FAS (full analysis set) 分析和 PP (per-protocol) 分析, 意向性分析人群 (ITT) 将包括所有参加随机并至少接受一次访视 的受试者。该人群将基于随机治疗,该人群为主要人群并用于进行有效性分析。

符合方案人群 (PP) 将包括所有至少随机并接受一次访视且严格遵循研究方案的受试者。 数据库建立前,报告分析计划中将规定严重违背方案的受试者从PP 人群中排除。PP 人群只对 临床有效率提供支持分析。如果 PP 人群达到了 ITT 人群的 95%以上,则不必进行 PP 人群的分 析。

安全性人群(SAF)将包括所有参加随机并至少接受一次访视的受试者,如果参加随机的 人群与实际接受治疗的人群不一致,则安全性分析人群将基于实际接受治疗的人群。

各指标将在意向性分析人群和符合方案人群均进行分析。

根据瘢痕大小进行分层:分为两层,10-50cm2与50-200cm2,在统计分析时,采用 Mantel-Haenszel 分层分析法评估确定混杂变量分层,然后计算各层优势比值,进行各层优势 比齐性检验。如果齐性,则报告公共优势比,根据公共优势比与未调整优势比的大小关系, 判断混杂方向。否则,分别报告不同层的优势比。

# 9.8 试验对象的随机方法

本研究采用随机分组方法,于每次术前实时短信联系统计学专家,由统计学专家利用 SAS 软件包编程产生的随机号决定入组受试者的组别, 其随机信息由统计学专家保存, 并短信实 时告知研究者受试者所随机组别。

# 10. 研究用物品

下列物品将提供给研究单位和研究者:

(1) 研究方案; (2) 知情同意书; (3) CRF表; (4) 研究者手册(5) 试验中心档案; 研究者在收到以上物品时, 需要在签收单上签字和注明日期。

# 11. 伦理学

# 11.1 研究者的责任

研究者有责任保证临床试验严格遵从试验方案,中国 GCP 指南和相关法规的要求。

- (1) 选择有资格和经验的研究单位和研究人员;
- (2) 在研究开始前利用讲座和文字材料等向研究人员详细介绍研究方案的内容,并共同对可能发生的问题制定解决方案;
- (3) 对所有填写了知情同意书并筛选合格进入试验的受试者,均须认真、详细记录病例记录表中的任何项目,不得空项、漏项(无记录的空格划横线);
  - (4) 病例记录表中所有数据需与受试者病历数据核对,保证无误;
- (5) 病例记录表作为原始数据,做任何更正时只能划线,旁注改后数据,并有研究者签姓 名首字母缩写标注日期;
  - (6) 由监查员定期核查数据的完整性和准确性;
- (7) 如果发现数据有疑问,应及时和研究人员沟通并进行确认或修正;统计阶段对数据进行盲态核查。如存在偏差,由研究人员进行确认或修正。

#### 12.4 手术操作培训

为保证各个分中心能各自独立进行手术操作,在项目开始前,将按 SOP 内容进行培训,并且定期监查,以达到同质性。本项目的各个分中心均与我们医院建立了医联体,此前已经进行了相关的培训,在项目开始前,将对各个分中心的手术操作者进行培训考试,合格后才能正式开始临床试验。

#### 12.5 监查

### 12.5.1监查的目的

确保临床试验严格按方案和有关法规进行,保障数据的完整性、可靠性及多中心数据的一致性,同时协调试验进度的统一性。

## 12.5.2监查的内容

监查员定期到临床研究单位,监查和报告试验的进行情况,监查员有权核对与本研究有关的所有受试者的原始资料。监查内容主要包括:受试者是否符合入组标准;病例报告表(CRF)的填写是否及时、准确、完整、可信;受试者用药的方法、剂量是否符合方案要求;所有不良事件是否都记录在 CRF 表中;同时保证所有错误或遗漏得以改正,并经研究者签名和注明日期。

如果在临床试验过程中,出现与本研究有关或无关的严重不良事件或死亡病例(包括化疗相关性死亡),经管医生或所在医院立即采取适当的处理措施。

# 12.6 研究结束/中止:

#### 12.6.1研究结束

试验中最后一名受试者随访结束后,研究者应通知中山大学,此时可视为研究结束。按中山大学规定,本项目应在 10 年内完成。

#### 12.6.2研究中止

牵头单位研究者保留在任何时候结束试验或中止某一研究点的权利。原因包括但不限于:

- 1) 研究者不能遵守试验方案:
  - 2) 研究者无法招募到足够的受试者;
  - 3) 安全方面的考虑:
  - 4) 有足够的证据证明缺乏疗效。

#### 12.7 稽查:

监察员或主要研究者定期进行稽查,稽查本试验所有的研究记录,包括原始文件,并和 CRF 表对比。稽查前会通知研究单位作适当的准备。药品管理相关机构可能进行类似的检查。 在这种情况下,研究者应当立即通知研究单位。

#### 13. 研究进度

10年共完成 226 例受试者临床研究。

试验启动日期: 2018年12月

试验结束日期: 2028年12月

其中,符合入组条件的受试者约占病例的 30%,预计有 10%的符合条件的受试者拒绝进入试验,进入试验的病例中预计在 6 月的随访期内约有 10%的失访率,根据本课题组每年收治病例情况,预计需要 10 年时间完成 226 例病例收集。

#### 14. 创新性及特色

- 1、自体瘢痕真皮支架,节经医疗资源:首次运用自体瘢痕真皮支架原位移植于创面上,相比较传统的昂贵的脱细胞异体真皮支架,有效减轻了患者负担,并且,更利于真皮支架的成活。
- **2、结构与功能双重修复**:实现自体基底细胞具有促进植皮成活的功能,有望恢复皮肤的附属结构。
  - 3、缓解皮源不足: 自体、快速。
  - 4、供皮区:基于损伤控制的供皮区。

#### 附件:

#### 附件 1: VAS 疼痛评分

共 0 分-10 分: 0 分: 无痛; 3 分以下: 有轻微的疼痛,患者能忍受; 4 分-6 分:患者疼痛并影响睡眠,尚能忍受; 7 分-10 分:患者有渐强烈的疼痛,疼痛难忍。

#### 附件 2: 温哥华瘢痕量表

色泽(M): 0 皮肤颜色与身体其他部分比较近似正常, 1 色泽较浅, 2 混合色泽, 3 色泽较深

血管分布(V): 0 正常肤色与身体其他部分近似 1 肤色偏粉红 2 肤色偏红 3 肤色呈紫色

厚度(H): 0 正常 1 大于 0 至 1mm 2 大于 1 至 2mm 3 大于 2 至 4mm 4 大于 4mm 柔软度(P): 0 正常 1 柔软的(在最少阻力下皮肤能变形的) 2 柔顺的(在压力下能变形的)

3 硬的(不能变形的,移动呈块状,对压力有阻力) 4 弯曲(组织如绳状,瘢痕伸展时会退缩)5 挛缩(瘢痕永久性缩短引致残废与扭曲)

最高分15分,最低分0分,分数越高说明瘢痕越重,反之,则轻.



### 研究流程表

| | 筛选期 | 入组 | 手术研究治疗期 | | | 随访评估 | |
|---|---|---|---|---|---|---|---|
| 访视窗口 | 访视 1 | 访视<br>2 | 访视3 | 访视 4 | 访视 5 | 访视 6 | 访视 7 |
| 评估/程序 | 术前-<br>10天内 | 手术当天 | 术后第1<br>周±1天 | 术后第2<br>周士3天 | 术后1个<br>月±5天 | 术后3个<br>月±7天 | 术后6个<br>月±7天 |
| 签署知情同意书 | X | | | | | 1100 | |
| 审查入选/排除标准 | X | | | | | | |
| 医学史(包括创伤史) | X | i and the second | | | | | |
| 血清妊娠试验2 | X | | | | | | |
| 进行创面检查和记录<br>生命体征 | X | х | х | Х | X | Х | X |
| 审查既往/联合用药 | X | X | X | Х | | | |
| 采集安全性试验血样<br>和尿样 | X | | | | | | |
| 随机分组 | | X | 121-1-1-105 | | | | |
| 审查不良事件4 | х | | X(术后研究治疗期<br>每日) | | | | |
| 监测术后研究治疗术<br>区的情况 <sup>5</sup> | | X | X(术后研究治疗期<br>每日) | | х | X | х |
| 给予研究治疗 | | X (据<br>分组<br>行植<br>皮术) | | | | | |
| 记录研究治疗信息 | | X | X | X | | - | |
| 审查体征和提供植皮<br>区描述 | Х | х | X | X | X | Х | X |

- 1 在术后第2周进行停止手术研究治疗期访视,在术后第2周进行植皮成活率评估。
- 2 在所有有生育能力的女性患者中进行血清妊娠试验。在研究期间还必须使用适当的避孕方法。
- 3 继续监测严重的和非严重的不良事件,直至术后3个月。必须进行末次安全性随访。
- 4 在手术后研究治疗期内每日监测创面情况。

6、 预期目标、年度计划及考核指标(前三年具体,后续年度可以简略) 预期目标

预期在前三年内实现超过40%的受试者入组,提高患者愈后质量,减少医疗费用

年度计划

争取在 7-8 年内完成受试者入组,在剩余研究时期内,进行数据整理,分析,撰写论文,在国际权威杂志上发表相关成果。

考核指标: 受试者入组数 病例报告表 四、项目实施年限及年度计划安排

| 项目实施总年限 | | 10 年 |
|---|---|---|
| | | 年度计划安排 |
| 时间进度 | | 阶段目标主要内容及成果 |
| 20 18年 12月-2019年 3 | 月 | 召开研究启动会议<br>组织课题组成员系统学习及培训<br>依照 CRF 内容建立电子数据库以便数据统计分析 |
| 20 19 年 4 月-2022 年 12 | 2月 | 按方案开展临床试验,筛选和入组受试者,完成治疗研究和随访<br>召开中期交流评价(每年评价分析一次试验方案的安全性并针对临床实践运作中的问题进行讨论分析,提出相应的解决办法)<br>完成 CRF 表和电子数据库<br>每半年由监察员进行监察及稽查 |
| 2023年1月-2026年1 | 2 月 | 继续按方案开展临床试验,筛选和入组受试者,完成治疗研究和随访,在此阶段结束前完成最后一例受试者的入组完成 CRF 表和电子数据库 召开中期交流评价(每年评价分析一次试验方案的安全性并针对临床实践运作中的问题进行讨论分析,提出相应的解决办法) 每半年由监察员进行监察及稽查 |
| 2027年1月-2028年1 | 2 月 | 按方案完成病例临床资料随访<br>完成 CRF 表和电子数据库<br>整理分析数据,撰写发表论文 |
| 20 年 月-20 年 | 月 | |
| 20 年 月-20 年 | 三月 | |
| 20 年 月-20 年 | 三 月 | |
| 20 年 月-20 年 | 手 月 | |

## 五、项目承担单位提供的技术及条件保障

(包括临床研究中心建设情况以及提供的人、财、物等支撑条件,该栏目由承担单位负责填写)

中山大学附属第一医院拥有 28 个临床重点专科,烧伤科是中华医学会烧伤外科分会**全国主任委员单位**,广东省内本专业唯一的"国家临床重点专科",广东省"临床重点专科","五个一科教兴医"工程重点学科,是华南地区知名科室,学术气氛浓厚,临床病例数多。能够保障课题组成员每年的工作时间,保障课题所需的临床标本量。

承担单位保证提供配套经费。

章) 【【】烟气量。【圆草一医院

年 月 日

# 六、项目经费支出总预算

单位:万元(保留两位小数)

| | 和 | 目名称 | | | 合计 | | 学校<br>经费 | 单位<br>配套 | | 自筹<br>经费 |
|---|---|---|---|---|---|---|---|---|---|---|
| 合 计 | | | | | 180 | | 90 | 90 | | |
| 1. 禾 | 斗研业务 | 费 | | | | | | | | |
| (1) 材料费 | | | | | 46 | | 23 | 23 | | |
| ( | (2) 差旅 | 费 | | | 13 | | 6. 5 | | 6.5 | |
| (3) 会议费 | | | | | 13 | | 6. 5 | | 6.5 | |
| | (4) 出版<br>以事务费 | 物/文献 | /信息传 | 播/知 | 13 | | 6.5 | 6.5 | | |
| | | (化验加] | Γ.费 | | 23 | | 11.5 | 11.5 | | |
| 2. 仪器设备费(不得购置大型仪器<br>设备) | | | | | | | | | | |
| (1) 购置设备费 | | | | | 4 | | 2 | 2 | | |
| (2) 设备改造与租赁费 | | | | | 0 | | 0 | 0 | | |
| <ol> <li>国际合作与交流费(不超过 10%)</li> <li>专家咨询费</li> <li>人员劳务费(不超过 30%)</li> </ol> | | | | | 16 | | 8 | | 8 | 3 |
| | | | | | | | 1 | 1 | | |
| | | | | | 46 | | 23 | 23 | | |
| 6. 其它(临床观察随访费等可归入 | | | | 4 | | 2 | | 2 | | |
| 此本 | 年份 | 2018年 | 2019年 | 2020年 | 2021年 | 2022年 | 2023年 | 2024年 | 2025年 | 2026年 |
| 年度 | 学校经. 费 | 10 万元 | 10 万元 | 10 万元 | 10 万元 | 10 万元 | 10 万元 | 10万元 | 10万元 | 10 万万 |
| 预 算 | 单位配套 | 10 万元 | 10 万元 | 10 万元 | 10 万元 | 10万元 | 10万元 | 10 万元 | 10万元 | 10 万万 |
| 31 | 白筹经<br>费 | | | | | | | | | |

### 对学校预算的详细说明(测算依据):

- 1. 科研业务费
- (1) 材料费: 电子数据库 RedCap 平台租借费用 0.3万/年, 手术所需耗材,器械
- (2) 差旅费: 参加国内会议 10 人次, 注册费 1000-元, 住宿 500 元/天, 会期 2-3 天, 往返车票/机票共 2500 元
- (3) 会议费:组织召开会议每年一次,会期 1-2 天,场地费约 5000 元/次,住宿费、伙食费等约 600 元/人天
- (4) 出版物/文献/信息传播/知识产权事务费:发表中文文章约4000元/篇,英文文章润饰费约1.0万元/篇
- (5) 测试化验加工费: 手术耗材加工, 检测等费用约 3000 元/次
- 2. 仪器设备费 (不得购置大型仪器设备)
- (1) 购置设备及维护检修费:购置手术器械,相机等现有设备的维护检修费约500元/次
- (2) 设备改造与租赁费
- 3. 国际合作与交流费: 需定期与国外专家进行互访交流,接收最新的资讯
- 4. 专家咨询费: 付统计专家分析、咨询费用
- 5. 人员劳务费: 聘请科研助手,参与研究生劳务费等,每月800元,每年平均工作8-10个月,科研助手需长期协助项目。
- 6. 其它(临床观察随访费等可归入此科目):每位受试者信件、电话及部分家访等费用,受试者回院复查交通补贴费(提高随访率之必须)(每例 200 元,共 226 例)

### 对单位配套的详细说明(测算依据):

- 1. 科研业务费
- (1) 材料费: 电子数据库 RedCap 平台租借费用 0.3万/年, 手术所需耗材, 器械
- (2) 差旅费: 参加国内会议 10 人次, 注册费 1000 元, 住宿 500 元/天, 会期 2-3 天, 往返车票/机票共 2500 元
- (3) 会议费:组织召开会议每年一次,会期 1-2 天,场地费约 5000 元/次,住宿费、工作餐等费用约 600 元/人天
- (4) 出版物/文献/信息传播/知识产权事务费:发表中文文章约4000元/篇,英文文章润饰费约1.0万元/篇
- (5) 测试化验加工费: 手术耗材加工, 检测等费用约 3000 元/次
- 2. 仪器设备费 (不得购置大型仪器设备)
- (1) 购置设备及维护检修费: 购置手术器械, 相机等现有设备维护检修费 200 元/次
- (2) 设备改造与租赁费
- 3. 国际合作与交流费: 需定期与国外专家进行互访交流,接收最新的资讯
- 4. 专家咨询费: 付统计专家分析、咨询费用
- 5. 人员劳务费: 聘请科研助手,参与研究生劳务费等,每月800元,每年平均工作8-10个月,科研助手需长期协助项目。
- 6. 其它(临床观察随访费等可归入此科目):每位受试者信件、电话及部分家访等费用,受试者回院复查交通补贴费(提高随访率之必须)(每例 200 元,共 226 例)

对自筹经费预算的详细说明(测算依据):

# 七、2019年度项目经费支出预算

单位: 万元 (保留两位小数)

| 利日石物 | | 学校 | 单位 | 位小数<br><b>自筹</b> |
|-------------------------|------|-------|-------|------------------|
| 科目名称 | 合计 | 经费 | 配套 | 经费 |
| 合 计 | 20 | 10 | 10 | |
| 1. 科研业务费 | | | | |
| (1) 材料费 | 4.8 | 2. 4 | 2. 4 | |
| (2) 差旅费 | 1.5 | 0. 75 | 0.75 | |
| (3) 会议费 | 1.5 | 0. 75 | 0.75 | |
| (4) 出版物/文献/信息传播/知识产权事务费 | 1.5 | 0. 75 | 0. 75 | |
| (5)测试化验加工费 | 2. 5 | 1. 25 | 1. 25 | |
| 2.仪器设备费(不得购置大型仪器设备) | | | | |
| (1) 购置设备费 | 0. 5 | 0. 25 | 0. 25 | |
| (2)设备改造与租赁费 | 0 | 0 | 0 | |
| 3. 国际合作与交流费(不超过 10%) | 2. 0 | 1 | 1 | |
| 4. 专家咨询费 | 0. 2 | 0.1 | 0. 1 | |
| 5. 人员劳务费(不超过 30%) | 5 | 2. 5 | 2. 5 | |
| 6. 其它(临床观察随访费等可归入此科目) | 0. 5 | 0. 25 | 0. 25 | |

对经费预算的其他说明:

# 经费支出预算填写说明:

- 1、 经费支出预算包括总经费支出预算和年度经费支出预算。
- 2、总经费支出预算中:
- (1) 常规项目: 学校经费、单位配套经费各 10 万元/年(具体按照项目批复的年限填写), 年度支出预算本次只预算 2018 年经费支出, 其中学校经费、单位配套经费各 10 万元, 以后逐年进行预算。
- (2) 培育项目: 学校经费、单位配套经费各 10 万元, 年度支出预算本次只预算 2018 年经费支出, 其中学校经费、单位配套经费各 5 万元。
- 3、如有合作单位,对方的经费预算请在合作协议中明确,注意要符合高校基本科研业务费经费管理要求。
- 4、经费用途及要求具体如下:
- (1) 科研业务费: 材料费、会议差旅费、论文发表费、成果与知识产权事务相 关费用、测试化验加工费等。
- (2) 仪器设备费:不得购置 40 万以上的大型仪器设备。
- (3) 国际合作与交流费: 不超过10%。
- (4) 人员劳务费: 用于直接参加项目研究的研究生、聘请人员等劳务费用,不得超过资助经费的 30%。
- (5) 专家咨询费: 标准参照国家和学校的相关规定执行。
- (6)管理费:根据高校基本业务费管理办法,高校基本业务费资助项目不得提取管理费,因此不在预算中列出。
- (7) 上述费用之外的其它支出,在申请预算时单独列示,单独核定。如临床病例观察随访费(用于支付入选临床病例医疗费用中与项目研究相关的检查、治疗费用及追踪随访费用)可以归入此科目。

# 八、项目组成员中统计学专家意见

(需附流行病或统计学专家签订的合作协议,复印件即可)

统计方法设计合理。

统计学专家签名 杂年表

2019年3月1日

# 九、承担单位伦理委员会意见

(需附伦理委员会批件)

伦理委员会成员签名

年 月 日

### 十、附件

1、合作单位研究协议书(如有合作单位请提供)

(合作协议中应明确承担单位与合作单位之间研究任务分工、经费分配、知识产权归属与分

- 享。请承担单位及合作单位的项目负责人、法人代表签名并加盖单位公章。)
- 2、伦理委员会批件。
- 3、流行病或统计学专家签订的合作协议(复印件即可)。
- 4、自筹资金承诺函。

# 十一、任务书签订各方意见

# 中山大学(甲方)

# 同意立项

负责人 (签名):



### 项目负责人(乙方)

项目负责人(签名)

年 月 日

# 项目承担单位(丙方)

申请者所在单位领导的审查意见与保证

已对任务书内容进行了审核:

- (1) 保证对研究计划实施所需的人力、物力和工作时间等条件给予支持
- (2) 承诺配套经费 10 万元/年度
- (3) 督促项目负责人按规定及时报送有关报表和材料

财务负责人(签名):